CLINICAL TRIAL: NCT03875807
Title: The Effect of Knee Flexion Angle for Graft Fixation During Single-Bundle Anterior Cruciate Ligament Reconstruction - A Multicentre, Patient and Assessor Blinded, Stratified, Two-arm Parallel Group Superiority Trial
Brief Title: The Effect of Knee Flexion Angle for Graft Fixation During Single-Bundle Anterior Cruciate Ligament Reconstruction
Acronym: KFA-FIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Arthroscopy Association of North America (Other)
Responsible Party: Principal Investigator, Dr. Jas Chahal, Orthopaedic Surgeon, Principle Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0006-B
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL; ACL reconstruction; Knee Flexion Angle; Bone Patellar Tendon Bone
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: A Multicentre, Pragmatic, Patient and Assessor Blinded, Stratified, Two-arm Parallel (1:1) Group Superiority Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients, assessors, and data analysts will be blinded in regards to treatment status at all times. Surgeons cannot be blinded given the nature of the intervention. We do not anticipate any circumstance in which unmasking of the data management team, or data analysts will be required, or permissible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0 degree Knee Flexion Angle ACLR (Active Comparator): At the time of surgery, tunnel position and surgical technique will be standardized for transtibial and anteromedial portal ACLR. Individuals randomized to this arm intra-operatively to undergo fixation of the ACL graft on the tibial side at a KFA of 0 degrees as measured by a sterile goniometer. Grafts will be tensioned according to the maximum surgeon-applied tension at the designated KFA. After surgery, patients will be treated with a standardized accelerated physical therapy protocol
  Interventions: Procedure: ACLR done at 0 degrees KFA
- 30 degree Knee Flexion Angle ACLR (Active Comparator): At the time of surgery, tunnel position and surgical technique will be standardized for transtibial and anteromedial portal ACLR. Individuals randomized to this arm intra-operatively to undergo fixation of the ACL graft on the tibial side at a KFA of 30 degrees as measured by a sterile goniometer. Grafts will be tensioned according to the maximum surgeon-applied tension at the designated KFA. After surgery, patients will be treated with a standardized accelerated physical therapy protocol
  Interventions: Procedure: ACLR done at 30 degrees KFA

INTERVENTIONS:
Procedure: ACLR done at 0 degrees KFA — Patients randomized to this arm will undergo the following intervention: Anterior Cruciate Ligament Reconstruction (ACLR) done at 0 degrees knee angle flexion (KFA)
  Arms: 0 degree Knee Flexion Angle ACLR
Procedure: ACLR done at 30 degrees KFA — Patients randomized to this arm will undergo the following intervention: Anterior Cruciate Ligament Reconstruction (ACLR) done at 30 degrees knee angle flexion (KFA)
  Arms: 30 degree Knee Flexion Angle ACLR

SUMMARY:
The overall aim of this study is to determine the effect of the knee flexion angle (KFA) of either 0 degrees, or 30 degrees (measured by sterile goniometer) during anterior cruciate ligament (ACL) fixation on postoperative outcomes following single-bundle ACL reconstruction with bone patellar tendon bone (BPTB) autograft. The specific aims of the current study include determining the effect of the knee flexion angle on 1) patient-reported outcomes; 2) postoperative extension loss; 3) antero-posterior (AP) knee stability; 4) rate of re-operation.

DETAILED DESCRIPTION:
At the present time, there is no consensus about the position of the knee during tensioning anterior cruciate ligament (ACL) graft fixation at the time of reconstruction, although it can be assumed to be one of the key factors for successful ACL reconstruction (ACLR). In studies that have investigated transtibial ACLR, it was suggested that 20 degrees is the ideal KFA to optimize graft force and the relative Antero-Posterior (AP) tibiofemoral relationship, while several other authors have advocated fixation in full extension to avoid overconstraining the knee. In the setting of anatomic ACLR, it has been reported that the tensioning of the graft at 30 degrees of knee flexion was associated with loss of knee extension when the anatomic femoral tunnel was chosen. Previous studies have performed gait analysis during walking in 24 patients with ACLR with hamstring autograft where graft fixation was performed at 25 degrees of knee flexion. In these study, the trans tibial (TT) technique resulted in significantly greater anterior femoral translation than healthy controls during the swing phase and excessive tibial internal rotation (IR) was found at midstance. In knees repaired with the anteromedial portal (AMP) technique, subjects were significantly less extended (5 degrees) compared with controls in late stance phase. While the AMP technique has the potential to improve overall joint stability, patients were shown to have increased difficulty with knee extension. It has also been demonstrated that since the anteromedial (AM) and posterolateral (PL) bundles of the ACL are at their longest in knee extension, the best angle for fixation would be near full extension. The aforementioned studies support the concept that anatomic ACL has an increased likelihood of anisometry and as a result the chosen KFA for fixation becomes increasingly important.

The lack of consensus regarding the optimal KFA in ACLR is reflected in the practice patterns of surgeons. A survey of Canadian Orthopaedic Surgeons demonstrated that 40% of surgeons fix the ACL at a 30 degree KFA while 30% perform fixation in full extension. The purpose of this study is to conduct a randomized controlled trial to determine if the KFA during ACLR graft fixation has an effect on postoperative outcomes. Patients undergoing single bundle BPTB ACLR will be randomized to have the surgical repair done with a KFA of either 0 degrees, or 30 degrees (measured by sterile goniometer) during anterior cruciate ligament (ACL) fixation. Patients will be followed for 24 months post surgery, with a number of qualitative patient surveys and clinical measurements being collected at 3, 6, 12 and 24 months post op, with changes being compared to baseline survey response and clinical measurement scores.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 16 years old with an isolated anterior cruciate ligament injury as diagnosed by clinical examination and MRI
* No pre-existing arthritis as defined by the Kellgren-Lawrence radiographic rating system
* Patients treated with an initial period of rehabilitation to eliminate swelling, optimize quadriceps strength and restore range of motion
* Surgical management with a transtibial or anteromedial portal single-bundle ACLR with bone patella tendon bone (BPTB) autograft by a fellowship-trained sports medicine surgeon.
* Provision of Informed Consent

Exclusion Criteria:

* Acute ACL injuries that have not undergone an initial period of physical therapy in order to restore the aforementioned parameters
* Associated grade III injury to the MCL (medial opening >10mm at 30 degrees of knee flexion or any medial opening in extension);
* Presence of a PCL or posterolateral corner injury
* Lack of informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Completed 24 months post ACL repair at 0 or 30 degrees flexion
  The KOOS questionnaire consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Completed 3, 6 and 12 months post ACL repair at 0 or 30 degrees flexion
  The KOOS questionnaire consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Marx Activity Score questionnaire | Completed at 3, 6, 12, 24 months post ACL repair at 0 or 30 degrees flexion
  The Marx Scale is a validated survey for orthopaedics that consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year.
  It is designed to be completed in less than one minute. The questionnaire is focused on actions that may be affected by disorders of the knee.
Loss of Extension on Operative Knee | Extension is measured at 3, 6, 12 and 24 months post ACL repair
  Extension loss versus contralateral knee measured clinically in degrees with a goniometer
Side to side differences in Anterior Posterior joint stability as measured by the KT-1000 Arthrometer | KT-1000 measurements are recorded at 3, 6,12 and 24 months post ACL repair
  The KT-1000 knee arthrometer (KT-1000) is an objective instrument to measure anterior tibial motion relative to the femur for anterior cruciate ligament (ACL) reconstruction. Measurements are captured on both the operative and non operative knee, and recorded at 0 degrees and 25 degrees flexion with a support placed under the knee for the latter measurement
Rate of Reoperation | Patients are followed for 24 months post initial ACL surgery to capture any instances of reoperation on the affected knee
  Rate of reoperation is recorded from date of original surgery to 24 months post original ACL repair, reoperations captured include retear of ACL, and any meniscus related tears.

CONTACTS AND LOCATIONS:
Overall Officials: Jas Chahal, MD, MSc, MBA, Principal Investigator — Women's College Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chahal J, Whelan DB, Hoit G, Theodoropoulos J, Ajrawat P, Betsch M, Docter S, Dwyer T. Anterior Cruciate Ligament Patellar Tendon Autograft Fixation at 0 degrees Versus 30 degrees Results in Improved Activity Scores and a Greater Proportion of Patients Achieving the Minimal Clinical Important Difference For Knee Injury and Osteoarthritis Outcome Score Pain: A Randomized Controlled Trial. Arthroscopy. 2022 Jun;38(6):1969-1977. doi: 10.1016/j.arthro.2021.12.018. Epub 2021 Dec 22. PMID 34952186